CLINICAL TRIAL: NCT03098173
Title: A Multi-center, Randomized Controlled Trial Comparing Early Versus Elective Colonoscopy in Outpatients With Acute Lower Gastrointestinal Bleeding
Brief Title: Comparing Early Versus Elective Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokyo University (Other)
Responsible Party: Principal Investigator, Atsuo Yamada, Department of Gastroenterology, Tokyo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2015034-11Y; UMIN000021129 (Other: University hospital Medical Information Network)
Record Dates: First submitted 2017-03-26; First posted 2017-03-31 (Actual); Results first posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-10

CONDITIONS: Acute Lower Gastrointestinal Bleeding
Keywords: Early colonoscopy; Stigmata of recent hemorrhage; Rebleeding

STUDY DESIGN:
Intervention Model Description: Parallel, randomized, superiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early colonoscopy (Experimental): Performance of prepared colonoscopy within 24 h of arrival
  Interventions: Procedure: Early colonoscopy
- Elective colonoscopy (Active Comparator): Performance of prepared colonoscopy between 24 and 96 h after arrival
  Interventions: Procedure: Elective colonoscopy

INTERVENTIONS:
Procedure: Early colonoscopy — Performance of prepared colonoscopy within 24 h of arrival
  Arms: Early colonoscopy
Procedure: Elective colonoscopy — Performance of prepared colonoscopy between 24 and 96 h after arrival
  Arms: Elective colonoscopy

SUMMARY:
This multi-center, randomized controlled trial study is planned to include 162 outpatients with onset of acute lower gastrointestinal bleeding to compare the rate of identification of stigmata of recent hemorrhage (SRH), and other clinical outcomes, including the 30-day rebleeding rate, between 'early' colonoscopy and 'elective' colonoscopy.

DETAILED DESCRIPTION:
All patients will receive early colonoscopy or elective colonoscopy, but they do so by different timing.

Early colonoscopy will be performed within 24 h of the initial visit. Elective colonoscopy will be performed between 24 and 96 h after the initial visit.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥ 20 years, presenting with moderate-to-severe hematochezia or melena within 24 h of arrival, defined as (i) more than three occurrences of hematochezia within 8 h, (ii) hemorrhagic shock, or (iii) requiring transfusion.
2. Provision of signed and dated informed consent form.
3. Stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Patients with hematemesis, black vomiting, or melena.
2. Patients with upper gastrointestinal bleeding, diagnosed by nasogastric tube or upper endoscopy.
3. Patients who have impossible consumed the oral bowel preparation solution.
4. Patients who have undergone computed tomography.
5. Patients who have been diagnosed with peptic ulcer diseases within the previous 10 days.
6. Ulcerative colitis or Crohn's disease patients.
7. Patients who have undergone abdominal surgery within the previous 10 days.
8. Patients who have undergone polypectomy, endoscopic mucosal resection, or endoscopic submucosal dissection of the lower gastrointestinal tract within the previous 10 days.
9. Patients with suspected perforation or peritonitis.
10. Patients with suspected intestinal obstruction.
11. Patients with hemorrhagic shock refractory to infusion or blood transfusion.
12. Patients who have undergone total colectomy.
13. Patients with suspected disseminated intravascular coagulation.
14. Patients with end-stage malignant disease.
15. Patients with severe cardiac failure.
16. Patients with active thrombosis.
17. Patients with severe respiratory failure.
18. Pregnant patients.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2016-01-29 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2019-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Atsuo Yamada, MD, Study Director — Tokyo University
Locations (15):
- Japan (15):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Hirosaki University Hospital, Hirosaki-shi, Aomori
  - National Center for Global Health and Medicine kohnodai hospital, Ichikawa-shi, Chiba
  - Fukui prefectural hospital, Fukui-shi, Fukui
  - National Hospital Organization Hakodate Hospital, Hakodate-shi, Hokkaido
  - Otaru Ekisaikai Hospital, Otaru-shi, Hokkaido
  - Tonan Hospital, Sapporo, Hokkaido
  - Ishikawa prefectural central hospital, Kanazawa, Ishikawa-ken
  - Nagasaki Harbor Medical Center City Hospital, Nagasaki, Nagasaki
  - Japan Community Healthcare Organization Osaka Hospital, Fukushima-shi, Osaka
  - Toyonaka Municipal Hospital, Toyonaka-shi, Osaka
  - The University of Tokyo, Bunkyo-ku, Tokyo
  - St. Luke's International Hospital, Chuo-ku, Tokyo
  - National Center for Global Health and Medicine center hospital, Shinjuku-ku, Tokyo
  - Shuto General Hospital, Yanai-shi, Yamaguchi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Niikura R, Nagata N, Doyama H, Ota R, Ishii N, Mabe K, Nishida T, Hikichi T, Sumiyama K, Nishikawa J, Uraoka T, Kiyotoki S, Fujishiro M, Koike K. Current state of practice for colonic diverticular bleeding in 37 hospitals in Japan: A multicenter questionnaire study. World J Gastrointest Endosc. 2016 Dec 16;8(20):785-794. doi: 10.4253/wjge.v8.i20.785. PMID 28042393
- [Derived] Niikura R, Nagata N, Yamada A, Honda T, Hasatani K, Ishii N, Shiratori Y, Doyama H, Nishida T, Sumiyoshi T, Fujita T, Kiyotoki S, Yada T, Yamamoto K, Shinozaki T, Takata M, Mikami T, Mabe K, Hara K, Fujishiro M, Koike K. Efficacy and Safety of Early vs Elective Colonoscopy for Acute Lower Gastrointestinal Bleeding. Gastroenterology. 2020 Jan;158(1):168-175.e6. doi: 10.1053/j.gastro.2019.09.010. Epub 2019 Sep 26. PMID 31563627
- [Derived] Niikura R, Nagata N, Yamada A, Doyama H, Shiratori Y, Nishida T, Kiyotoki S, Yada T, Fujita T, Sumiyoshi T, Hasatani K, Mikami T, Honda T, Mabe K, Hara K, Yamamoto K, Takeda M, Takata M, Tanaka M, Shinozaki T, Fujishiro M, Koike K. A multicenter, randomized controlled trial comparing the identification rate of stigmata of recent hemorrhage and rebleeding rate between early and elective colonoscopy in outpatient-onset acute lower gastrointestinal bleeding: study protocol for a randomized controlled trial. Trials. 2018 Apr 3;19(1):214. doi: 10.1186/s13063-018-2558-y. PMID 29615078

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Elective Colonoscopy | Early Colonoscopy
Started | 81 | 81
Completed | 80 | 79
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Colonoscopy | Elective Colonoscopy | Total
Number analyzed (Participants) | 79 | 80 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (12.8) | 71.9 (12.3) | 70.3 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 26 | 53
  Male | 52 | 54 | 106
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 79 | 80 | 159
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 23.0 (3.3) | 23.9 (4.1) | 23.5 (3.7)
Previous lower GI bleeding [Count of Participants; unit: Participants] | 28 | 30 | 58
Ischemic heart disease [Count of Participants; unit: Participants] | 12 | 18 | 30
Chronic obstructive pulmonary disease [Count of Participants; unit: Participants] | 3 | 0 | 3
Peptic ulcer [Count of Participants; unit: Participants] | 6 | 2 | 8
Liver cirrhosis [Count of Participants; unit: Participants] | 1 | 2 | 3
Diabetes mellitus [Count of Participants; unit: Participants] | 11 | 16 | 27
Chronic heart failure [Count of Participants; unit: Participants] | 4 | 5 | 9
Cerebrovascular disease [Count of Participants; unit: Participants] | 11 | 15 | 26
Dementia [Count of Participants; unit: Participants] | 0 | 2 | 2
Collagen disease [Count of Participants; unit: Participants] | 4 | 5 | 9
Chronic kidney disease [Count of Participants; unit: Participants] | 8 | 11 | 19
Leukemia [Count of Participants; unit: Participants] | 0 | 1 | 1
Malignant lymphoma [Count of Participants; unit: Participants] | 2 | 0 | 2
Solid cancer [Count of Participants; unit: Participants] | 7 | 12 | 19
Low-dose aspirin [Count of Participants; unit: Participants] | 16 | 22 | 38
Thienopyridine [Count of Participants; unit: Participants] | 7 | 6 | 13
Cilostazol [Count of Participants; unit: Participants] | 5 | 2 | 7
Other antiplatelet drugs [Count of Participants; unit: Participants] | 5 | 3 | 8
Warfarin [Count of Participants; unit: Participants] | 4 | 6 | 10
Direct oral anticoagulants [Count of Participants; unit: Participants] | 3 | 7 | 10
NSAIDs [Count of Participants; unit: Participants] | 14 | 16 | 30
Hemodynamic instability [Count of Participants; unit: Participants] | 4 | 1 | 5
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 11.4 (2.7) | 11.3 (2.3) | 11.3 (2.5)
Upper GI endoscopy before colonoscopy [Count of Participants; unit: Participants] | 2 | 1 | 3
Expert endoscopist [Count of Participants; unit: Participants] | 48 | 48 | 96
Cecal insertion [Count of Participants; unit: Participants] | 77 | 77 | 154
Cecal insertion time [Mean (Standard Deviation); unit: minutes] | 9.6 (19.2) | 9.0 (6.5) | 9.3 (6.5)
Total procedure time [Mean (Standard Deviation); unit: minutes] | 35.8 (19.2) | 31.3 (15.1) | 33.6 (17.4)
Bleeding source [Number; unit: participants]
  Diverticular bleeding (definite) | 10 | 16 | 26
  Diverticular bleeding (presumptive) | 37 | 36 | 73
  Colorectal cancer | 3 | 2 | 5
  Ischemic colitis | 9 | 5 | 14
  Infectious colitis | 1 | 0 | 1
  Radiation colitis | 1 | 0 | 1
  Colonic ulcer | 0 | 2 | 2
  Hemorrhoid | 1 | 2 | 3
  Other | 7 | 4 | 11
  Unknown | 13 | 13 | 26
  Upper GI bleeding | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Stigmata of Recent Hemorrhage (SRH) Identification Rate
Description: Stigmata of Recent Hemorrhage (SRH) based on colonoscopic visualization of lesions, such as diverticulosis, tumor, ulcer, hemorrhoid, angioectasia, and polyps exhibiting active bleeding, a visible vessel, or an adherent clot.
Time Frame: 0-4 day
Population: The primary analysis included a modified intention-to-treat population, excluding the following patients from the genuine intention-to-treat analysis set: 1) those who did not satisfy the enrollment criteria after randomization; 2) those who provided no post-randomization data on primary outcome; and 3) those who did not undergo colonoscopy
Measure: Count of Participants; unit: Participants
Arm/Group | Early Colonoscopy | Elective Colonoscopy
Number analyzed (Participants) | 79 | 80
Participants | 17 | 17

2. Secondary Outcome: Success Rate of Endoscopic Treatment; Number of Participants Achieving Hemostasis With Endoscopic Treatment
Description: Success rate will be defined as the number achieving hemostasis per total number of attempts at endoscopic hemostasis during colonoscopy examination.
Time Frame: 0-4 day
Population: Success rate of endoscopic treatment was defined as achievement of hemostasis (early for 15 patients and elective for 15 patients).
Measure: Count of Participants; unit: Participants
Arm/Group | Early Colonoscopy | Elective Colonoscopy
Number analyzed (Participants) | 15 | 15
Participants | 14 | 15

3. Secondary Outcome: Need for Additional Endoscopic Examinations
Description: Additional endoscopic examinations will be defined as examinations to achieve hemostasis.
Time Frame: 0-34 day
Measure: Count of Participants; unit: Participants
Arm/Group | Elective Colonoscopy | Early Colonoscopy
Number analyzed (Participants) | 79 | 80
Participants | 31 | 23

4. Secondary Outcome: Need for Interventional Radiology
Description: It will be defined as radiology intervention to achieve hemostasis.
Time Frame: 0-34 day
Measure: Count of Participants; unit: Participants
Arm/Group | Early Colonoscopy | Elective Colonoscopy
Number analyzed (Participants) | 79 | 80
Participants | 1 | 0

5. Secondary Outcome: Need for Surgery
Description: It will be defined as surgery to achieve hemostasis.
Time Frame: 0-34 day
Measure: Count of Participants; unit: Participants
Arm/Group | Early Colonoscopy | Elective Colonoscopy
Number analyzed (Participants) | 79 | 80
Participants | 0 | 0

6. Secondary Outcome: Thirty-day Rebleeding Rates
Description: Rebleeding will be defined as significant fresh blood loss after an initial colonoscopy with any of the following criteria:
  i) Hemorrhagic shock, including cold sweat, nausea, syncope, or systolic blood pressure ≤ 90 mmHg.
  ii) Need for transfusion, according to the guidelines of the Ministry of Health, Labour, and Welfare.
  iii) Further colonoscopy identifies blood pooling, or iv) SRH in the lower gastrointestinal tract. v) Contrast-enhanced CT identifies extravasation in the colorectal region. However, these examinations will not be performed routinely if rebleeding occurs in the study period.
Time Frame: 30 day
Population: Rebleeding,thrombotic events, and mortality were evaluated for patients who approximately met the 30-day follow-up criteria (early colonoscopy for 72 patients and elective colonoscopy for 75 patients).
Measure: Count of Participants; unit: Participants
Arm/Group | Early Colonoscopy | Elective Colonoscopy
Number analyzed (Participants) | 72 | 75
Participants | 11 | 5

7. Secondary Outcome: Need for Transfusion During Hospitalization
Description: It will be defined as the numbers of patients who will need transfusion.
Time Frame: During hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | Early Colonoscopy | Elective Colonoscopy
Number analyzed (Participants) | 79 | 80
Participants | 30 | 26

8. Secondary Outcome: Length of Stay
Description: It will be defined as length of stay to cure acute lower gastrointestinal bleeding.
Time Frame: 0-34 day
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Early Colonoscopy | Elective Colonoscopy
Number analyzed (Participants) | 79 | 80
days | 7.1 (5.7) | 7.6 (6.0)

9. Secondary Outcome: Number of Participants With Thirty-day Thrombosis Events
Description: Thrombosis events will include acute coronary syndromes, including angina pectoris and myocardial infarction, stroke, including cerebrovascular infarction, cerebral hemorrhage, and transient ischemic attacks, deep vein thrombosis, and pulmonary embolism.
Time Frame: 30 day
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Early Colonoscopy | Elective Colonoscopy
Number analyzed (Participants) | 72 | 75
Participants | 1 | 0

10. Secondary Outcome: Number of Participants With Thirty-day Death Events
Description: Number of Participants with Thirty-day death Events from enrollment
Time Frame: 30 day
Measure: Count of Participants; unit: Participants
Arm/Group | Early Colonoscopy | Elective Colonoscopy
Number analyzed (Participants) | 79 | 80
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Preparation-related Adverse Events
Description: Preparation-related adverse events will include nausea, vomiting, abdominal pain, volume overload, aspiration pneumonia, hemorrhagic shock, exacerbation bleeding, and ileus
Time Frame: 0-4 day
Measure: Count of Participants; unit: Participants
Arm/Group | Early Colonoscopy | Elective Colonoscopy
Number analyzed (Participants) | 79 | 80
Participants | 36 | 28

12. Secondary Outcome: Number of Participants With Colonoscopy-related Adverse Events
Description: Colonoscopy-related adverse events will include hemorrhagic shock, and perforation.
Time Frame: 0-4 day
Measure: Count of Participants; unit: Participants
Arm/Group | Early Colonoscopy | Elective Colonoscopy
Number analyzed (Participants) | 79 | 80
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 30 day
Description: Data will be entered into a web-based EDC system by trial investigators or site investigators.
Arm/Group | Early Colonoscopy | Elective Colonoscopy
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/80
Serious Adverse Events (participants affected / at risk) | 2/79 | 0/80
Other Adverse Events (participants affected / at risk) | 9/79 | 8/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Colonoscopy (N=79) | Elective Colonoscopy (N=80)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0
Bacterial cellulitis (Infections and infestations) | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early Colonoscopy (N=79) | Elective Colonoscopy (N=80)
Hypoxemia (General disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Upper respiratory inflammation (Infections and infestations) | 1 | 0
Pseudogout (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute prostatitis (Renal and urinary disorders) | 1 | 0
Vagal reflex (Nervous system disorders) | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Pyrexia (Infections and infestations) | 2 | 2
Arthritis pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Abdominal bloating (Gastrointestinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Non blinding

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT03098173/Prot_SAP_000.pdf